CLINICAL TRIAL: NCT00187239
Title: Reduce Ventricular Pacing in Dual Chamber Implantable Cardioverter Defibrillators Using AutoIntrinsic Conduction Search (REDUCE Study)
Brief Title: Reduce Ventricular Pacing in Dual Chamber Implantable Cardioverter Defibrillators Using AutoIntrinsic Conduction Search Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Director, Scientific Studies, St. Jude Medical
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRD292
Record Dates: First submitted 2005-09-10; First posted 2005-09-16 (Estimated); Last update posted 2019-02-04 (Actual); Status verified 2019-02

CONDITIONS: Arrhythmia
Keywords: ICDs; Ventricular pacing; Patient has been implanted with a dual chamber SJM ICD with AICS for 1 month (± 2 weeks).; At the time of enrollment, patient is paced in the RV ≤25% of the time as determined by the device diagnostics.; Patient is medically stable.
MeSH Terms: conditions — Arrhythmias, Cardiac

ARMS (2):
- AICS On (Active Comparator): Patients in this arm have Autointrinsic conduction search programmed ON.
  Interventions: Device: Autointrinsic Conduction Search Algorithm
- AICS Off (No Intervention): Patients assigned to this arm do not have Autointrinsic Conduction Search programmed on.

INTERVENTIONS:
Device: Autointrinsic Conduction Search Algorithm — Autointrinsic conduction search is programmed on in those patients randomized to AICS ON.
  Arms: AICS On

SUMMARY:
The purpose of this study is to determine if patients implanted with a St. Jude Medical (SJM) implantable cardioverter defibrillator (ICD) will benefit by using AutoIntrinsic Conduction Search (AICS) rather than only a programmed AV/PV delay. This study will compare the two methods of programming with respect to intrinsic activity.

ELIGIBILITY:
Inclusion Criteria:

* Patient has been implanted with a dual chamber SJM ICD with AICS for 1 month (± 2 weeks).
* At the time of enrollment, patient is paced in the right ventricle (RV) ≤25% of the time as determined by the device diagnostics.
* Patient is medically stable.

Exclusion Criteria:

* Patient has evidence of atrioventricular (AV) block (first, second or third degree) such that ventricular pacing would be required as part of the patient's routine management
* Patient is unable to comply with the follow-up visits due to geographical, psychological, or any other reasons.
* Patient is younger than 18 years of age.
* Patient is pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 157 (Actual)
Dates: Start 2005-07; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
The primary endpoint is the percentage of intrinsic ventricular events. | 3 months

SECONDARY OUTCOMES:
Number of atrial tachycardia (AT), atrial fibrillation (AF), ventricular tachycardia (VT), and ventricular fibrillation (VF) episodes | 3 months
Frequency of inappropriate ICD therapy during AT/AF | 3 months
Frequency of appropriate ICD therapy for VT/VF | 3 months
Study related adverse events | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Zaffer Syed, MS, Study Director — Abbott Medical Devices
Locations (1):
- AtlantiCare Regional Medical Center, Pomona, New Jersey, United States